CLINICAL TRIAL: NCT06055803
Title: The Heart Health After Cancer Treatment (HEART-ACT): A Pilot Study of a Multi-disciplinary Health Behavior Intervention in People With a History of Breast Cancer to Reduce Heart Disease Risk After Cancer Treatment.
Brief Title: Heart Health After Cancer Treatment (HEART-ACT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 228014; NCI-2023-07108 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Health Behavioral Program; Cardiac Health
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Behavior Program (Experimental): Each participant will have an individualized assessment with plan and goals set at the program intake visit. Program components will include: Physical Activity, Nutrition, Emotional Well-being, Cardiovascular Risk, Survivorship, and other items individualized to the participant as needed (e.g., tobacco cessation). The 12-week program will alternate between group and individual sessions each week. Individualized plans will be reviewed every two weeks at the participant individual sessions.
  Interventions: Behavioral: Intake Session; Behavioral: Individual Sessions; Behavioral: Group Sessions; Behavioral: Graduation; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Intake Session — Each of the program components will have an individualized assessment with plan and goals set at the program intake visit.
Behavioral: Individual Sessions — Individual sessions will occur in person or virtual every other week during the 12-week intervention with a health promotion specialist (nurse or exercise physiologist). These sessions will include review of progress towards goals, update exercise prescription, make plan for the next two weeks.
Behavioral: Group Sessions — Group sessions for wellness and education will be delivered by medical multi-disciplinary staff in person or virtual every other week during the 12-week intervention.
Behavioral: Graduation — At the conclusion of the 12-week intervention, there will be a graduation session to honor the participant's achievement and establish a plan for maintenance after the intervention
Behavioral: Exercise — Participants will exercise as part of individual and group sessions. Participants will also be asked to exercise on their own, with a goal of working up to meeting US Physical Activity guidelines (150 minutes per week of moderate to vigorous exercise + 2 episodes of strength training).

SUMMARY:
This is a pilot study testing multi-disciplinary health behavior intervention in breast cancer survivors who have been treated at Zuckerberg San Francisco General (ZSFG).

DETAILED DESCRIPTION:
OBJECTIVES:

1. Evaluating feasibility and acceptability of the program.
2. Evaluating the effects of the program on health outcomes including change in exercise capacity, change in quality of life, change in risk factors, and adverse events.
3. Evaluating changes in patient-reported measures.

OUTLINE:

Participants with a history of breast cancer who receive care at Zuckerberg San Francisco General Hospital (ZSFG) will receive the intervention which is comprised of a 12-week multi-disciplinary health behavior program. Each participant will have an individualized assessment, goal and plan for each component of the program. Follow-up for outcomes will occur at 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Diagnosis of breast cancer
* Treated with curative intent
* Able to communicate in English, Spanish, or Cantonese
* Able to consent for self
* Receive care at Zuckerberg San Francisco General Hospital

Exclusion Criteria:

* Chemotherapy, radiation, or surgery planned in next 3 months
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with analyzable data for change in 6 Minute Walk Distance (6MWD) | Baseline to 12 months
  6MWD measures the distance walked over 6 minutes. The farther a person can walk indicates better exercise tolerance and mobility. The changes in distance will be compared at baseline and 12 months. We will measure the proportion of participants with analyzable 6MWD data.
Proportion of participants with analyzable data for change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health - Mental Scale | Baseline to 12 months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health. We will calculate the change in the score between baseline and 12 months. The proportion of participants who can have a score measured will be calculated.
Proportion of participants with analyzable data for change in PROMIS Global Health - Physical Health Scale | Baseline to 12 months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health. We will calculate the change in the score between baseline and 12 months.

SECONDARY OUTCOMES:
Net Promoter Score | 3 Months
  The Net Promoter Score asks the participant to report how likely they are to recommend this health behavior program to another breast cancer survivor on a scale of 1 (Very Unlikely) to 10 (Very Likely). The Score is calculated as the percent of respondents who are "promoters" reporting a 9 or 10 minus the percent of responders who are "detractors" reporting a 1-6. The score can range from -100 to 100, with 100 being the best score.
Net Promoter Score | 6 Months
  The Net Promoter Score asks the participant to report how likely they are to recommend this health behavior program to another breast cancer survivor on a scale of 1 (Very Unlikely) to 10 (Very Likely). The Score is calculated as the percent of respondents who are "promoters" reporting a 9 or 10 minus the percent of responders who are "detractors" reporting a 1-6. The score can range from -100 to 100, with 100 being the best score.
Net Promoter Score | 12 Months
  The Net Promoter Score asks the participant to report how likely they are to recommend this health behavior program to another breast cancer survivor on a scale of 1 (Very Unlikely) to 10 (Very Likely). The Score is calculated as the percent of respondents who are "promoters" reporting a 9 or 10 minus the percent of responders who are "detractors" reporting a 1-6. The score can range from -100 to 100, with 100 being the best score.
Change in 6MWD | Baseline and 12 Months
  6MWD measures the distance walked over 6 minutes. The farther a person can walk indicates better exercise tolerance and mobility. The changes in distance will be compared at baseline and 12 months.
Change in 6MWD | Baseline and 6 Months
  6MWD measures the distance walked over 6 minutes. The farther a person can walk indicates better exercise tolerance and mobility. The changes in distance will be compared at baseline and 6 months.
Change in 6MWD | Baseline and 3 Months
  6MWD measures the distance walked over 6 minutes. The farther a person can walk indicates better exercise tolerance and mobility. The changes in distance will be compared at baseline and 3 months.
Change in PROMIS Global Health - Mental Scale | Baseline and 12 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health. We will calculate the change in the score between baseline and 12 months.
Change in PROMIS Global Health - Mental Scale | Baseline and 6 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health. We will calculate the change in the score between baseline and 6 months.
Change in PROMIS Global Health - Mental Scale | Baseline and 3 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The mental health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better mental health. We will calculate the change in the score between baseline and 3 months.
Change in PROMIS Global Health - Physical Scale | Baseline and 12 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health. We will calculate the change in the score between baseline and 12 months.
Change in PROMIS Global Health - Physical Scale | Baseline and 6 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health. We will calculate the change in the score between baseline and 6 months.
Change in PROMIS Global Health - Physical Scale | Baseline and 3 Months
  The PROMIS Global Health 10 questionnaire is a self-assessed questionnaire that asks participants to respond to 10 questions. The physical health subscale consists of four questions with a raw score between 4 and 20 that is converted to a standardized T-score. Higher scores represent better physical health. We will calculate the change in the score between baseline and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Beatty, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Analytic and community advisory board members will be provided with de-identified study data.